CLINICAL TRIAL: NCT01622218
Title: The Impact of Medical Clowning on Pain and Stress Level in Pediatric Patients Undergoing Hernia Repair Surgery LAUGH Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Nitza Heiman Newman, MD, Principle Investigator, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sor007112clit
Record Dates: First submitted 2012-05-30; First posted 2012-06-19 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Umbilical Hernia; Inguinal Hernia
Keywords: Medical clown
MeSH Terms: conditions — Hernia, Umbilical; Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Clown (Experimental): Presence of clowns on child's postoperative pain levels, anxiety levels of the child and the accompanying parent and the effect of the intervention on the total consumption of analgesics and on the post- surgery inflammatory markers.
  Interventions: Behavioral: Medical Clown
- Control (No Intervention): Assessment of child's postoperative pain levels, anxiety levels of the child and the accompanying parent and the effect on the total consumption of analgesics and on the post- surgery inflammatory markers.

INTERVENTIONS:
Behavioral: Medical Clown — Presence of clowns on child's postoperative pain levels, anxiety levels of the child and the accompanying parent and the effect of the intervention on the total consumption of analgesics and on the post- surgery inflammatory markers
  Arms: Medical Clown

SUMMARY:
The purpose of our study to quantitatively examine the stress levels prior to surgery and the use of analgesics post surgery in both children and their parents following a preoperative intervention with a medical clown compared to children that were not exposed to this intervention.

ELIGIBILITY:
Inclusion Criteria:

* ages 4-10 years old
* undergoing elective umbilical or inguinal hernia repair surgery
* ASA Physical Status = 1

Exclusion Criteria:

* None

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Children: WBS (Wong Baker Faces Pain Rating Scale) | 24 hours
  measure at 4 time points (repeated measures) - at admission, discharge, 12 and 24 hours.

SECONDARY OUTCOMES:
Use of analgesics | During the 24 hours following the surgery
  Total dose of analgesics over 24 periods per kg.
Cytokines levels | End of precedure, before waking up
  Cytokined levels at the end of the surgery (end of precedure, before waking up)(IL-1b, IL-2,IL-6, IL-8, IL-10,TNF-α and VEGF)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Assuta Medical Center, Beersheba